CLINICAL TRIAL: NCT03988140
Title: Could the Apico-coronal Position of the Implant Influence the Peri-implant Parameters in Mandibular Edentulous Type 2 Diabetics Rehabilitated With Implant-retained Overdentures? A Split-mouth RCT With 24-months Follow up.
Brief Title: Apico-coronal Position of the Implant in Edentulous Diabetics With Implant-retained Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Fernanda Vieira Ribeiro, Principal Investigator, Paulista University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: apico-coronal position
Record Dates: First submitted 2019-05-30; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus; Dental Implants
Keywords: dental prosthesis; biological markers; dental implants
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This study was designed as a prospective, split-mouth, randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implant placed at supra crestal level (SL) (Experimental): Implants were placed at supra crestal level (SL)
  Interventions: Device: Dental Implant Placement and subsequent prosthetic reabilithation
- Implant placed at crestal level (CL). (Other): Implants were placed at crestal level (CL)
  Interventions: Device: Dental Implant Placement and subsequent prosthetic reabilithation

INTERVENTIONS:
Device: Dental Implant Placement and subsequent prosthetic reabilithation — Surgeries to dental implant placement were performed. All patients received 3.5 mm diameter dental implants - surface blasted with TiO2 particles and machined collar of 1mm - in the interforaminal region of the mandible. The surgical sequence followed the protocol described by the implant company.A two stages protocol was used and the prostheses were placed at 4 months.The prosthetic retention system used in rehabilitation with overdentures was the O'ring and the capture of this component was done directly in the patient's mouth. After 7 and 14 days, the patients returned to occlusal adjustments and verification of prosthetic adaptation. The prostheses were made entirely of acrylic resin without metallic reinforcement and the antagonist of the patients were total edentulous and rehabilitated with muco-supported prostheses.

SUMMARY:
Diabetes Mellitus (DM) is a recognized factor affecting implant complication rates, including peri-implantitis and peri-implant bone loss, and the apico-coronal position of implants seems interfere on the conditions of peri-implant tissues. However, the influence of the vertical implant position in type 2 diabetics (T2DM) is unclear. This split-mouth randomized controlled trial evaluated the impact of implants of machined-collar placed at crestal level or supracrestally in T2DM rehabilitated with implant-retained overdentures on the clinical, tomographic and immunoinflammatory peri-implant outcomes after implant loading.

DETAILED DESCRIPTION:
Considering the outcomes achieved with implants with machined-collar inserted supracrestally, it would be relevant to investigate whether this therapeutic strategy could be considered as a more effective approach in the rehabilitation with dental implants of individuals with type 2 DM, since these patients may be more disposed to peri-implant changes, both from the point of view of marginal bone remodeling as related to local variations in immunoinflammatory response. Thus, the propose of this split-mouth randomized controlled trial was to compare the impact of crestal level or supracrestally implant platform in T2DM rehabilitated with implant-retained overdentures on the clinical, tomographic and immunoinflammatory peri-implant outcomes after implant loading.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria included: patients aged between 50 and 80 years old, 2) totally edentulous in the mandible with previous mandibular dentures for at least 6 months and indicated for rehabilitation with overdenture, 3) patients with diabetes had to have had T2DM, diagnosed by a physician, for at least the past 5 years. Such individuals were either under a dietary regimen and/or were using oral hypoglycaemic agents (metformin or glybenclamin).

Exclusion Criteria:

* Exclusion criteria were: 1) pregnancy, 2) lactation, 3) current smoking or ex-smokers, 4) other systemic conditions that could affect bone metabolism (e.g., immunologic disorders), 5) use of anti-inflammatory, immunosuppressive and anti-resorptive medications, 6) patients that required bone grafts before or concomitantly with implant surgery and 7) a history of previous regenerative procedures in the area designated for implant therapy. Patients with major complications of DM (i.e., cardiovascular and peripheral vascular diseases [ulcers, gangrene, and amputation], neuropathy, and nephropathy) were also excluded.

Ages: 59 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline Peri-implant Probing Depth (PPD) at 24 months. | (baseline) and at 6, 12 and 24 months
  distance from the bottom of the peri-implant pocket (PPD) to the mucosal margin (MM) measured by a calibrated examiner in millimeter using a Periodontal probing

SECONDARY OUTCOMES:
Mucosal Margin (MM) | (baseline) and at 6, 12 and 24 months
  distance from the implant platform to the peri-implant margin (CL group) and distance from the machined collar maintained supracrestally to the peri-implant margin (SL group) measured by a calibrated examiner in millimeter using a Periodontal probing
Clinical attachment level (CAL) | (baseline) and at 6, 12 and 24 months
  calculated by adding PPD and MM measured by a calibrated examiner in millimeter using a Periodontal probing
Modified Bleeding on Probing | (baseline) and at 6, 12 and 24 months
  dichotomous index of bleeding during probing around implants measured by a calibrated examiner using a Periodontal probing. Data were presented as percentage.
Modified Plaque Index | (baseline) and at 6, 12 and 24 months
  dichotomous modified plaque index along the mucosal margin around implants measured by a calibrated examiner using a Periodontal probing. Data were presented as percentage.
Crest Height Bone Marginal Peri-implant | (baseline) and at 6, 12 and 24 months
  linear measurement in millimeter obtained by a parallel line to the implant surface from the implant platform to bone crestal (mesial, distal, buccal and lingually) in the sagittal and coronal slices each 2 mm using Cone Beam Computed Tomography (CBCT) scans
Markers on peri-implant crevicular fluid | (baseline) and at 6, 12 and 24 months
  The levels of Imunoinflammatory mediators: interferon (IFN)-gama, interleukin (IL)-10, IL-17, IL-33, IL-21, IL-4, IL-23, IL-6 and tumor necrosis factor (TNF)-α in the peri-implant crevicular fluid were determined using human plex and the multiplexing instrument. The mean concentration of each biomarker was calculated and expressed as pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Conte, Study Chair — Paulista U

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogurtsova K, da Rocha Fernandes JD, Huang Y, et al. IDF Diabetes Atlas: Global estimates for the prevalence of diabetes for 2015 and 2040. Diabetes Res Clin Pract. 2017; 128:40-50. GBD 2016 DALYs and HALE Collaborators. Global, regional, and national disability-adjusted life-years (DALYs) for 333 diseases and injuries and healthy life expectancy (HALE) for 195 countries and territories, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet, 390: 1260-1344. Kapur KK, Garrett NR, Hamada MO, et al. A randomized clinical trial comparing the efficacy of mandibular implant-supported overdentures and conventional dentures in diabetic patients. Part I: Methodology and clinical outcomes. J Prosthet Dent. 1998; 79: 555-569.
- [Derived] Conte A, Ghiraldini B, Denofrio PHF, Marcello-Machado RM, Correa MG, Pimentel SP, Casati MZ, Pecorari VGA, Cirano FR. Supracrestal implant placement improves peri-implant health in T2DM patients: A randomized clinical trial. J Dent. 2025 Oct;161:106002. doi: 10.1016/j.jdent.2025.106002. Epub 2025 Jul 25. PMID 40716558